CLINICAL TRIAL: NCT00317941
Title: The AVANTAGE Study - A Randomized, Multicenter, Phase IV, Open-label Prospective Study Comparing Injection Site Reaction and Injection Site Pain in Patients With Relapsing Remitting Multiple Sclerosis (RRMS) or After a First Demyelinating Event Suggestive of MS Newly Started on Interferon Beta-1b (Betaferon®) or Interferon Beta-1a (Rebif®).
Brief Title: Safety Study in Relapsing-remitting Multiple Sclerosis (RRMS) Patients Receiving Betaferon or Rebif
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Healthcare AG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 91489; 2005-005583-91 (EudraCT Number); 308084 (Other: company internal); Avantage (Other: company internal)
Record Dates: First submitted 2006-04-24; First posted 2006-04-25 (Estimated); Results first posted 2013-10-21 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2013-08

CONDITIONS: Relapsing-remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; RRMS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Interferon beta-1b; Interferon beta-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- IFNB-1b 250 mcg (Betaseron) via Betaject (Experimental): Interferon beta 1b ([IFNB-1b] Betaseron, BAY86-5046) 250 mcg (8 MIU) administered every other days by subcutaneous injection using Betaject
  Interventions: Drug: Betaferon/Betaseron
- IFNB-1b 250 mcg (Betaseron) via Betaject light (Experimental): Interferon beta 1b ([IFNB-1b] Betaseron, BAY86-5046) 250 mcg (8 MIU) administered every other days by subcutaneous injection using Betaject Light
  Interventions: Drug: Betaferon/Betaseron
- IFNB-1a 44 mcg (Rebif) via Rebiject II (Active Comparator): Interferon beta-1a ([IFNB-1a] Rebif) 44 mcg (12 MIU) three times per week by subcutaneous injection using Rebiject II
  Interventions: Drug: Rebif

INTERVENTIONS:
Drug: Betaferon/Betaseron — 250ug administrated with Betaject
  Arms: IFNB-1b 250 mcg (Betaseron) via Betaject
Drug: Rebif — 44ug administered with Rebiject II
  Arms: IFNB-1a 44 mcg (Rebif) via Rebiject II
Drug: Betaferon/Betaseron — 250ug administrated with Betaject light
  Arms: IFNB-1b 250 mcg (Betaseron) via Betaject light

SUMMARY:
The purpose of this study is to compare the injection site reaction and injection site pain after subcutaneous administration of either Betaferon 250µg or Rebif 44µg using different autoinjectors.

DETAILED DESCRIPTION:
Original French title of the study: Etude de phase IV, multicentrique, randomisée, ouverte, comparant les réactions et la douleur aux sites d'injection après administration sous-cutanée d'interféron β-1b (Betaferon®) ou interféron β-1a (Rebif®) pendant la période de trois mois d'initiation de la thérapie chez des patients atteints d'une forme récurrente/rémittente de sclérose en plaques.

The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer HealthCare AG, Germany. Bayer HealthCare AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Males or females
* Age >= 18 years old
* Patients after a first demyelinating event suggestive of MS (only for Betaferon) as well as patients with a definite diagnosis of RRMS (Betaferon et Rebif)
* First justified prescription of one interferon beta by subcutaneous route (as described in Summary of Product Characteristics [SmPC] of Betaferon or Rebif)
* Females of child-bearing potential must agree to practice adequate contraceptive methods over the duration of the study (not applicable for men)
* Patient can follow and comply with all study procedures of the trial protocol
* Laboratory evaluations (i.e., evaluation of hepatic enzyme gamma-GT, full blood count and differential white blood cell count [WBC]) must be available and the results must be normal.
* Written informed consent

Exclusion Criteria:

* Any contraindication to the prescription of Betaferon or Rebif, as described in the SmPC of products:

  * Pregnancy or lactation
  * Known hypersensitivity to natural or recombinant interferon beta, to mannitol, to human albumin or any other excipients used
  * History of severe depression or suicide attempt or current suicidal ideation.
  * Patient with decompensated liver disease
  * Epilepsy not adequately controlled by treatment
* Patient previously included in this study.
* Patient previously treated by sub-cutaneous route with either Betaferon or Rebif.
* Participation in any clinical trial within the past 30 days involving the investigational drug intake.
* Medical, psychiatric or other conditions that compromise the patient's ability to understand the patient information, to give informed consent, to comply with the trial protocol or to complete the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2006-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (56):
- France (56):
  - Aix-en-Provence
  - Alkirch
  - Annecy
  - Aurillac
  - Belfort
  - Blaye
  - Bordeaux
  - Boulogne-sur-Mer
  - Brest
  - Brive-la-Gaillarde
  - Carcassonne
  - Castelnau-le-Lez
  - ChamaliÃ¿res
  - Champigny-sur-Marne
  - Colmar
  - Corbeil Essones Cedex
  - CrÃ©teil
  - Dijon
  - Dreux
  - Dunkirk
  - Elbeuf
  - Évreux
  - Évry
  - La Seyne-sur-Mer
  - Le Mans
  - Libourne
  - Lille
  - Lomme
  - Lyon
  - Marseille
  - Montpellier
  - Nancy
  - Nantes
  - Nice
  - Nîmes
  - Paris
  - Pau
  - Perpignan
  - Poissy
  - Quimper
  - Reims
  - Rennes
  - Rouen
  - Rueil-Malmaison
  - Saint LÃ¿
  - Saint-Etienne
  - Saint-Herblain
  - Saint-Omer
  - Saint-Quentin
  - Strasbourg
  - Toulouse
  - Tourcoing
  - Trélazé
  - Vendôme
  - Vesoul
  - Vichy

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: IFNB-1b 250 Mcg (Betaseron) Via Betaject: Interferon beta 1b ([IFNB-1b] Betaseron, BAY86-5046) 250 mcg (8 MIU) administered every other days by subcutaneous injection using Betaject
- Group B: IFNB-1b 250 Mcg (Betaseron) Via Betaject Light: Interferon beta 1b ([IFNB-1b] Betaseron, BAY86-5046) 250 mcg (8 MIU) administered every other days by subcutaneous injection using Betaject Light
- Group C: IFNB-1a 44 Mcg (Rebif) Via Rebiject II: Interferon beta-1a ([IFNB-1a] Rebif) 44 mcg (12 MIU) three times per week by subcutaneous injection using Rebiject II
Period: Overall Study
Arm/Group | Group A: IFNB-1b 250 Mcg (Betaseron) Via Betaject | Group B: IFNB-1b 250 Mcg (Betaseron) Via Betaject Light | Group C: IFNB-1a 44 Mcg (Rebif) Via Rebiject II
Started | 73 | 79 | 68
Participants Received Treatment | 73 | 79 | 68
Fulfilled Requirement Safety Population | 73 | 77 | 65
Fulfilled Requirements PP Population | 66 | 76 | 63
Completed | 66 | 74 | 60
Not Completed | 7 | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- IFNB-1b 250 Mcg (Betaseron): Interferon beta 1b ([IFNB-1b] Betaseron, BAY86-5046) 250 mcg (8 MIU) administered every other days by subcutaneous injection using Betaject or Betaject Light
- Total: Total of all reporting groups
Arm/Group | IFNB-1b 250 Mcg (Betaseron) | IFNB-1a 44 Mcg (Rebif) Via Rebiject II | Total
Number analyzed (Participants) | 142 | 63 | 205
Age Continuous [Mean (Standard Deviation); unit: Years] | 39.2 (10.3) | 38.4 (10.5) | 38.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 47 | 153
  Male | 36 | 16 | 52
Number of relapses [Mean (Standard Deviation); unit: Relapses] | 2.2 (1.2) | 2.1 (1.0) | 2.1 (1.1)
Expanded disability status scale at screening (EDSS) [Mean (Standard Deviation); unit: Scores on a scale] — The EDSS scores range from 0.0 (normal) to 10.0 (dead). A score of 2 to 3 indicates minimal to moderate disability.
  Scores on a scale | 1.7 (1.2) | 1.9 (1.4) | 1.8 (1.3)
Time since diagnosis [Mean (Standard Deviation); unit: Years] | 3.3 (5.7) | 3.3 (6.7) | 3.3 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of the Sites Developing a Injection Site Reaction (ISR) Reported by Participants 24 Hours After Each Injection
Description: An injection site is seen as developing a reaction if the patient's score for this site is of a reaction intensity ≥ 1. Number of injection sites per month per participant analyzed
Time Frame: Up to 3 months assessed every 24 hours after each injection
Measure: Number; unit: Percentage of sites
Units Other Than Participants: injection sites per month per patient
Arm/Group | IFNB-1b 250 Mcg (Betaseron) | IFNB-1a 44 Mcg (Rebif) Via Rebiject II
Number analyzed (Participants) | 142 | 63
Number analyzed (injection sites per month per patient) | 16 | 16
Percentage of sites | 31 | 37

2. Primary Outcome: Percentage of Sites Developing a Injection Site Reaction (ISR) Reported by Participants 48 Hours After Each Injection
Description: as for outcome 1
Time Frame: Up to 3 months assessed every 48 hours after each injection
Measure: Number; unit: Percentage of sites
Units Other Than Participants: Injection sites per month per patient
Arm/Group | IFNB-1b 250 Mcg (Betaseron) | IFNB-1a 44 Mcg (Rebif) Via Rebiject II
Number analyzed (Participants) | 142 | 63
Number analyzed (Injection sites per month per patient) | 16 | 16
Percentage of sites | 27 | 41

3. Primary Outcome: Mean Scores of Reaction After Injection Reported by Participants
Description: Score range is: 0 - no abnormal reaction, 1 -erythema, 2-edema, 3-infiltration, 4-ulceration or necrosis
Time Frame: Up to 3 months assessed every 24 and 48 hours after injection
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: Injection sites per month per patient
Arm/Group | IFNB-1b 250 Mcg (Betaseron) | IFNB-1a 44 Mcg (Rebif) Via Rebiject II
Number analyzed (Participants) | 142 | 63
Number analyzed (Injection sites per month per patient) | 16 | 16
Scores on a scale | 0.368 (3.11) | 0.500 (3.45)

4. Other Pre Specified Outcome: Mean Scores of Reaction After Injection Reported by Patients Between Different Auto Injectors
Description: Score range is: 0 - no abnormal reaction, 1 -erythema, 2-edema, 3-infiltration, 4-ulceration or necrosis
Time Frame: Up to 3 months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: Injection sites per month per patient
Arm/Group | IFNB-1b 250 Mcg (Betaseron) Via Betaject | IFNB-1b 250 Mcg (Betaseron) Via Betaject Light | IFNB-1a 44 Mcg (Rebif) Via Rebiject II
Number analyzed (Participants) | 66 | 76 | 63
Number analyzed (Injection sites per month per patient) | 16 | 16 | 16
Scores on a scale | 0.372 (2.82) | 0.363 (3.34) | 0.5 (3.45)

5. Secondary Outcome: Percentage of Injection Sites With Pain Reported by Physicians
Time Frame: Up to 3 months
Measure: Number; unit: Percentage of sites
Units Other Than Participants: Injection sites per month per patient
Arm/Group | IFNB-1b 250 Mcg (Betaseron) | IFNB-1a 44 Mcg (Rebif) Via Rebiject II
Number analyzed (Participants) | 142 | 63
Number analyzed (Injection sites per month per patient) | 16 | 16
Percentage of sites | 6.2 | 5.2

6. Secondary Outcome: Percentage of Injection Sites Per Participant With Reaction Reported by Physicians
Time Frame: Up to 3 months
Measure: Number; unit: Percentage of ISR
Units Other Than Participants: Injection sites per month per patient
Arm/Group | IFNB-1b 250 Mcg (Betaseron) | IFNB-1a 44 Mcg (Rebif) Via Rebiject II
Number analyzed (Participants) | 142 | 63
Number analyzed (Injection sites per month per patient) | 16 | 16
Percentage of ISR | 14.1 | 18.6

7. Secondary Outcome: Percentage of Participants Without ISR Reported by Participants
Time Frame: Up to 3 months assessed every 24 hours after each injection
Measure: Number; unit: Percentage of participants
Arm/Group | IFNB-1b 250 Mcg (Betaseron) | IFNB-1a 44 Mcg (Rebif) Via Rebiject II
Number analyzed (Participants) | 142 | 63
Percentage of participants | 21.3 | 9.5

8. Secondary Outcome: Percentage of Sites Developing a Severe Reaction 24 Hours After Injection
Description: An ISR is considered as severe if the score reported by the patient is above 2 (at least one red skin) 0- no abnormal reaction, 1- erythema, 2-edema, 3- infiltration 4- ulceration or necrosis
Time Frame: Up to 3 months assessed every 24 hours after each injection
Measure: Number; unit: Percentage of sites
Units Other Than Participants: Injection sites per month per patient
Arm/Group | IFNB-1b 250 Mcg (Betaseron) | IFNB-1a 44 Mcg (Rebif) Via Rebiject II
Number analyzed (Participants) | 142 | 63
Number analyzed (Injection sites per month per patient) | 16 | 16
Percentage of sites | 6.1 | 8.45

9. Secondary Outcome: Percentage of Sites Developing a Severe Reaction 48 Hours After Injection
Description: as for outcome 8
Time Frame: Up to 3 months assessed every 48 hours after each injection
Measure: Number; unit: Percentage of sites
Units Other Than Participants: Injection sites per month per patient
Arm/Group | IFNB-1b 250 Mcg (Betaseron) | IFNB-1a 44 Mcg (Rebif) Via Rebiject II
Number analyzed (Participants) | 142 | 63
Number analyzed (Injection sites per month per patient) | 16 | 16
Percentage of sites | 4.97 | 8.76

10. Secondary Outcome: Percentage of Participants Without Pain Reported by Participants
Time Frame: Up to 3 months assessed 24 hours after each injection
Measure: Number; unit: Percentage of participants
Arm/Group | IFNB-1b 250 Mcg (Betaseron) | IFNB-1a 44 Mcg (Rebif) Via Rebiject II
Number analyzed (Participants) | 142 | 63
Percentage of participants | 5.6 | 17.7

11. Secondary Outcome: Percentage of Injection Sites Without Pain Reported by Physicians
Time Frame: Up to 3 months
Measure: Number; unit: Percentage of injection sites
Units Other Than Participants: Injection sites per month per patient
Arm/Group | IFNB-1b 250 Mcg (Betaseron) | IFNB-1a 44 Mcg (Rebif) Via Rebiject II
Number analyzed (Participants) | 142 | 63
Number analyzed (Injection sites per month per patient) | 16 | 16
Percentage of injection sites | 85.9 | 81.4

12. Secondary Outcome: Percentage of Injection Sites Without Pain Reported by Participants
Time Frame: Up to 3 months assessed 24 hours after each injection
Measure: Number; unit: Percentage of injection sites
Units Other Than Participants: Injection sites per month per patient
Arm/Group | IFNB-1b 250 Mcg (Betaseron) | IFNB-1a 44 Mcg (Rebif) Via Rebiject II
Number analyzed (Participants) | 142 | 63
Number analyzed (Injection sites per month per patient) | 16 | 16
Percentage of injection sites | 30.3 | 42.0

13. Secondary Outcome: Mean Pain Assessment Using Visual Analogue Scale (VAS) Reported by Participants Immediately After Injection
Description: Visual analogue scale was used to report the pain from 0 (no pain ) to 10 (maximal pain).
Time Frame: Immediately after injection
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | IFNB-1b 250 Mcg (Betaseron) Via Betaject | IFNB-1a 44 Mcg (Rebif) Via Rebiject II
Number analyzed (Participants) | 142 | 63
Scores on a scale | 1.1992 [0 to 8.6714] | 1.4502 [0 to 6.1636]

14. Secondary Outcome: Mean Pain Assessment Using Visual Analogue Scale (VAS) Reported by Participants 30 Minutes After Injection
Description: Visual analogue scale was used to report the pain from 0 (no pain ) to 10 (maximal pain).
Time Frame: 30 min after injection
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | IFNB-1b 250 Mcg (Betaseron) Via Betaject | IFNB-1a 44 Mcg (Rebif) Via Rebiject II
Number analyzed (Participants) | 142 | 63
Scores on a scale | 0.7046 [0 to 8.7429] | 0.8461 [0 to 6.8286]

15. Secondary Outcome: Mean Pain Assessment Using Visual Analogue Scale (VAS) Reported by Participants 1 Hour After Injection
Description: Visual analogue scale was used to report the pain from 0 (no pain ) to 10 (maximal pain).
Time Frame: 1h after injection
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | IFNB-1b 250 Mcg (Betaseron) Via Betaject | IFNB-1a 44 Mcg (Rebif) Via Rebiject II
Number analyzed (Participants) | 142 | 63
Scores on a scale | 0.5737 [0 to 8.5857] | 0.6666 [0 to 9.6]

16. Secondary Outcome: Mean Pain Assessment Using Visual Analogue Scale (VAS) Reported by Participants 24 Hours After Injection
Description: Visual analogue scale was used to report the pain from 0 (no pain ) to 10 (maximal pain).
Time Frame: 24h after injection
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | IFNB-1b 250 Mcg (Betaseron) Via Betaject | IFNB-1a 44 Mcg (Rebif) Via Rebiject II
Number analyzed (Participants) | 142 | 63
Scores on a scale | 0.6411 [0 to 8.8071] | 0.5811 [0 to 9.2333]

17. Secondary Outcome: Percentage of Sites Without Reaction 24 Hours After Injection Reported by Participants
Time Frame: Up to 3 months assessed every 24 hours after each injection
Measure: Number; unit: Percentage of sites
Units Other Than Participants: Injection sites per month per patient
Arm/Group | IFNB-1b 250 Mcg (Betaseron) | IFNB-1a 44 Mcg (Rebif) Via Rebiject II
Number analyzed (Participants) | 142 | 63
Number analyzed (Injection sites per month per patient) | 16 | 16
Percentage of sites | 62.2 | 63.0

18. Secondary Outcome: Percentage of Sites Without Reaction 48 Hours After Injection Reported by Participants
Description: if the patient score is missing, at the injection site, then the patient is not considered without or with developping reaction.
  An injection site is seen as developing no reaction if the patient's score for this site is of a reaction intensity = 0.
Time Frame: Up to 3 months assessed every 48 hours after each injection
Measure: Number; unit: Percentage of sites
Units Other Than Participants: Injection sites per month per patient
Arm/Group | IFNB-1b 250 Mcg (Betaseron) | IFNB-1a 44 Mcg (Rebif) Via Rebiject II
Number analyzed (Participants) | 142 | 63
Number analyzed (Injection sites per month per patient) | 16 | 16
Percentage of sites | 71.8 | 54.6

ADVERSE EVENTS:
Groups:
- IFNB-1b 250 Mcg (Betaseron): Interferon beta 1b ([IFNB-1b] Betaseron, BAY86-5046) 250 mcg (8 MIU) administered every other days by subcutaneous injection using Betaject or Betaject Light. Participants at risk from Group A and Group B in Participant flow.
- IFNB-1a 44 Mcg (Rebif) Via Rebiject II: Interferon beta-1a ([IFNB-1a] Rebif) 44 mcg (12 MIU) three times per week by subcutaneous injection using Rebiject II. Participants at risk from Group C in Participant flow.
Arm/Group | IFNB-1b 250 Mcg (Betaseron) | IFNB-1a 44 Mcg (Rebif) Via Rebiject II
Serious Adverse Events (participants affected / at risk) | 2/150 | 1/65
Other Adverse Events (participants affected / at risk) | 83/150 | 42/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IFNB-1b 250 Mcg (Betaseron) (N=150) | IFNB-1a 44 Mcg (Rebif) Via Rebiject II (N=65)
Lumbago (Musculoskeletal and connective tissue disorders) | 1 | 0
Cytolitic hepatitis (Hepatobiliary disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IFNB-1b 250 Mcg (Betaseron) (N=150) | IFNB-1a 44 Mcg (Rebif) Via Rebiject II (N=65)
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Palpitations (Cardiac disorders) | 4 | 0
Eye pain (Eye disorders) | 2 | 1
Ophtalmoplegia (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 2 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 6 | 5
Fatigue (General disorders) | 6 | 2
Feeling hot (General disorders) | 1 | 0
Hot flush (General disorders) | 1 | 1
Injection site inflammation (General disorders) | 1 | 0
Influenza like illness (General disorders) | 32 | 15
Injection site erythema (General disorders) | 3 | 1
Injection site oedema (General disorders) | 1 | 0
Injection site pain (General disorders) | 7 | 6
Injection site pruritus (General disorders) | 1 | 0
Irritability (General disorders) | 2 | 0
Malaise (General disorders) | 2 | 1
Pyrexia (General disorders) | 4 | 3
Hepatic pain (Hepatobiliary disorders) | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 2 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0
Furuncle (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 2 | 0
Alanine aminotransferase increase (Investigations) | 2 | 1
Aspartate aminotransferase increase (Investigations) | 1 | 0
Transaminase increase (Investigations) | 5 | 1
Decrease appetite (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemie (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbago (Musculoskeletal and connective tissue disorders) | 0 | 2
Chills (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 6 | 3
Hypoaesthesia (Nervous system disorders) | 3 | 0
Insomnia (Nervous system disorders) | 1 | 3
Multiple sclerosis relapse (Nervous system disorders) | 12 | 8
Paresthesia (Nervous system disorders) | 2 | 1
Somnolence (Nervous system disorders) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Depressed mood (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Parasomnia (Psychiatric disorders) | 0 | 1
Cystitis (Renal and urinary disorders) | 1 | 0
Urinary track infection (Renal and urinary disorders) | 2 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1
Ejaculation disorder (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 2 | 0
Hospitalization (Surgical and medical procedures) | 0 | 1
Dizziness (Vascular disorders) | 1 | 0
Hematoma (Vascular disorders) | 1 | 0
Venous insufficiency (Vascular disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Optic neuritis (Eye disorders) | 1 | 0
Initial insomnia (Nervous system disorders) | 1 | 0
Muscular weakness (Nervous system disorders) | 1 | 0
Motor dysfunction (Nervous system disorders) | 1 | 0
Pain (General disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
According the contract he signed, If results should have been edited, the Principal Investigators (PI) should have been obtained the agreement from the sponsor 90 days before the publication. The PI was not allowed to communicate within a public way the information on the study without having obtained the sponsor's agreement.